CLINICAL TRIAL: NCT03075449
Title: Real World Data Exploring the Practices of Primary Care Providers in the Managment of Male Lower Urinary Tract Symptoms
Brief Title: Real World Data on Management of Male LUTS
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.87
Record Dates: First submitted 2017-03-08; First posted 2017-03-09 (Actual); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study will describe the current medical care given to men who discuss their lower urinary tract symptoms with a HCP. It will document the primary reasons for the visit, the baseline characteristics of these men, the treatment received, and the practice patterns of specifically a primary care physician managing these patients.

ELIGIBILITY:
Inclusion criteria:

* Males, aged ≥18 years old.
* Having had discussion of urinary symptoms with their PCP between 15 days and 12 months prior to the date of the phone interview.
* Able to read, speak and understand English.
* Willing to provide informed consent for study participation, authorize the release of their previous 12-month medical records from their PCP for review and de-identified data entry by Mapi into an electronic study database.

Exclusion criteria:

* Reported during screening that they had had their first-ever discussion of urinary symptoms with PCP within the 14 days prior to the date of the phone interview.
* Participation in a clinical research study that evaluated urinary symptoms in the past 12 months.
* Self-reported history of colorectal, bladder or prostate cancer.
* Self-reported neurologic disorders that affect bladder function, e.g., neurogenic bladder disorders due to spinal cord injury/disease, multiple sclerosis, Parkinsons disease.
* Self-reported history of radiation therapy to the lower abdominal and/or pelvic region.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 527.87.10001 Boehringer Ingelheim Investigational Site, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A cross-sectional participant survey study combined with 12 months of retrospective data collection from participant's PCP medical records.
Groups:
- Participant Data Reported by Telephone Survey + Medical Record: Participant-reported data during the telephone survey and the medical record from the Primary Care Provider (PCP) from which medical data were abstracted by the medical data abstractor in the Management of Male Lower Urinary Tract Symptoms
Period: Overall Study
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Started | 170
Completed | 170
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The enrolled set contains all men who have met all study eligibility criteria and have returned the signed ICF. This includes meeting eligibility criteria according to medical records.
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 170

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Men Given a Drug Prescription for Their Urinary Symptoms, as Recorded in Their Medical Records
Description: The percentage of men who have been given at least one prescription medication for urinary symptoms.
  This included any medications prescribed by PCP for urinary symptoms according to medical records within 12 months prior to telephone survey as described below:
  1. Medications already prescribed by PCP for urinary symptoms prior to the 1st visit/contact for urinary symptoms within 12 months prior to telephone survey.
  2. Medications newly prescribed by PCP upon visit(s)/contact(s) for urinary symptoms within 12 months prior to telephone survey (i.e., medications prescribed for urinary symptoms on or after the 1st visit/contact).
  95% CI was calculated using clopper-pearson estimation method based on the exact binomial distribution.
Time Frame: 12 months
Population: Full Analysis Set (FAS): The FAS consists of all enrolled men whose PCP has provided their medical record with at least one urinary symptom recorded between 15 days and 12 months prior to telephone survey interview.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 84
Percentage of participants | 35.7 [25.6 to 46.9]

2. Secondary Outcome: The Percentage of Men Who Received a Medical Diagnosis for Their Urinary Symptoms, as Recorded in Their Medical Records.
Description: The percentage of men who received a medical diagnosis for their urinary symptoms, as recorded in their medical records.
  95% CI was calculated using clopper-pearson estimation method based on the exact binomial distribution.
Time Frame: 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 84
Percentage of participants | 79.8 [69.6 to 87.7]

3. Secondary Outcome: The Percentage of Men With a Diagnostic Testing Procedure Ordered or Performed Specifically for Their Urinary Symptoms.
Description: The percentage of men with a diagnostic testing procedure ordered or performed specifically for their urinary symptoms.
  95% CI was calculated using clopper-pearson estimation method based on the exact binomial distribution.
Time Frame: 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 84
Percentage of participants | 61.9 [50.7 to 72.3]

4. Secondary Outcome: The Percentage of Men Diagnosed With LUTS/BPH (Enlarged Prostate).
Description: The percentage of men diagnosed with lower urinary tract symptoms (LUTS)/benign prostatic hyperplasia (BPH) (enlarged prostate).
  95% CI was calculated using clopper-pearson estimation method based on the exact binomial distribution.
Time Frame: 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 84
Percentage of participants | 42.9 [32.1 to 54.1]

5. Secondary Outcome: The Percentage of Men Referred to a Urologist for Their Urinary Symptoms.
Description: The percentage of men referred to a urologist for their urinary symptoms.
  95% CI was calculated using clopper-pearson estimation method based on the exact binomial distribution.
Time Frame: 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 84
Percentage of participants | 48.8 [37.7 to 60.0]

6. Secondary Outcome: The Percentage of Men Given a Prescription for an Alpha-blocker for Their Urinary Symptoms.
Description: The percentage of men given a prescription for an alpha-blocker for their urinary symptoms.
  95% CI was calculated using clopper-pearson estimation method based on the exact binomial distribution.
Time Frame: 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 84
Percentage of participants | 26.2 [17.2 to 36.9]

7. Secondary Outcome: The Percentage of Men Given Repeat Prescriptions for Their Urinary Symptoms.
Description: The percentage of men given repeat prescriptions for their urinary symptoms.
  95% CI was calculated using clopper-pearson estimation method based on the exact binomial distribution.
Time Frame: 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 84
Percentage of participants | 33.3 [23.4 to 44.5]

8. Secondary Outcome: The Number of Urinary-symptom Related Visits to Their PCP During the 12 Month Period Prior to Telephone Survey Interview.
Description: The number of urinary-symptom related visits to their primary care provider (PCP) during the 12 month period prior to telephone survey interview.
Time Frame: 12 months
Population: FAS
Measure: Mean (Standard Deviation); unit: urinary symptom-related visits
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Number analyzed (Participants) | 84
urinary symptom-related visits | 1.8 (1.24)

ADVERSE EVENTS:
Description: No safety data was planned to be collected for this study thus adverse events are not reported.
Arm/Group | Participant Data Reported by Telephone Survey + Medical Record
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.